CLINICAL TRIAL: NCT04297150
Title: Identification of Clinical and Pharmacogenetic Factors Predictive of Response to New Oral Anticoagulants in the Treatment of Non-valvular Atrial Fibrillation.
Brief Title: Predictive Factors for Response to New Oral Anticoagulants in the Treatment of Non-valvular Atrial Fibrillation..
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Other Study IDs: SFC-NAC-2019-01
Record Dates: First submitted 2020-02-18; First posted 2020-03-05 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; edoxaban; Rivaroxaban; Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One tube of blood for DNA extration and genotyping. One tube of blood for plasma extraction and drug determination. One tube of blood for the determination of anticoagulant activity.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Patients that satisfy inclusion criteria: Patients who satisfy the inclusion criteria and sign the informed consent.
  Interventions: Drug: Apixaban; Drug: Edoxaban; Drug: Rivaroxaban; Drug: Dabigatran

INTERVENTIONS:
Drug: Apixaban — Drug indicated for the treatment of NVAF
  Other Names: Eliquis
Drug: Edoxaban — Drug indicated for the treatment of NVAF
  Other Names: Lixiana
Drug: Rivaroxaban — Drug indicated for the treatment of NVAF
  Other Names: Xarelto
Drug: Dabigatran — Drug indicated for the treatment of NVAF
  Other Names: Pradaxa

SUMMARY:
Post-authorization observational, prospective, follow-up study of a cohort of patients with non-valvular atrial fibrillation who are treated with direct oral anticoagulants (DOACs) to evaluate the clinical course (occurrence of stroke, major bleeding and mortality) and its correlation with clinical, pharmacokinetic (plasma concentrations), pharmacodynamic (haemostatic) and pharmacogenetic factors.

DETAILED DESCRIPTION:
Post-authorization observational, prospective, follow-up study of a cohort of patients with non-valvular atrial fibrillation treated with direct oral anticoagulants (dabigatran, rivaroxaban, apixaban and edoxaban) to assess the clinical course (occurrence of stroke, other ischemic or bleeding events and mortality) and its correlation with clinical, pharmacokinetic (plasma concentrations), pharmacodynamic (haemostatic) and pharmacogenetic factors.

Patient selection and follow-up will be performed in 6 public Spanish hospitals: Hospital Universitario de la Princesa, Hospital Universitario La Paz, Hospital Universitario Ramón y Cajal, Fundación Jiménez Díaz, Hospital Gómez Ulla (Madrid) and Hospital Universitario de Burgos (Burgos). To reduce variability, the determination of anticoagulant activity will be performed in the Hematology Service of the Hospital Universitario de Burgos and the measurement of plasma concentrations and genotyping of all patients in the Clinical Pharmacology Service of the Hospital Universitario de la Princesa.

Patients who are to receive or are receiving one of the four DOACs currently available in Spain will be informed about the characteristics of this study and will be asked to sign the consent form for their participation. The treatment or clinical management of these patients at each centre will not be modified. They will be asked three blood samples, coinciding with other tests that will be carried out to monitor their pathology (one blood sample for the study of the effect on coagulation, another for drug quantification in plasma and another for genetic studies) with the only requirement that they must have been treated with the drug for at least one week so that they have spent more than 5 half-lives and are in steady state. The samples will be extracted in the morning, before medication intake (trough concentrations).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women over 18 years of age
2. Patients with non-valvular atrial fibrillation (NVAF).
3. Patients who are going to receive or are receiving treatment with any of the DOACs (dabigatran, rivaroxaban, apixaban or edoxaban) for the prevention of stroke and systemic embolism in adult patients with NVAF, according to the drug label.
4. Patients who agree to participate in the study and give their written consent.

Exclusion Criteria:

1. Patients on treatment with other anticoagulants.
2. Patients suffering from a malignant or terminal disease whose life expectancy is less than 6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over 18 years of age with NVAF requiring anticoagulant treatment with a DOAC. The prescription of the treatment will be previous and independent to the inclusion of the patient in the study. Patients who will initiate treatment (which will only be evaluated prospectively) and patients already in treatment (which will also be evaluated retrospectively) will be included.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Major haemorrhages | Throughout the follow-up, i.e. for at least 15 months and up to 30.
  Occurrence of haemorrhages will be monitored throughout the follow-up, i.e. for at least 15 months and up to 30.

SECONDARY OUTCOMES:
Haemorragic stroke | Throughout the follow-up, i.e. for at least 15 months and up to 30.
  Occurrence of haemorragic stroke will be monitored throughout the follow-up i.e. for at least 15 months and up to 30..
Ischemic stroke | Throughout the follow-up, i.e. for at least 15 months and up to 30.
  Occurrence of ischemic stroke will be monitored throughout the follow-up i.e. for at least 15 months and up to 30..
Death | Throughout the follow-up, i.e. for at least 15 months and up to 30.
  All-cause mortality will be monitored throughout the follow-up i.e. for at least 15 months and up to 30..

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Gómez Ulla, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz:, Madrid
  - Hospital Universitario de La Paz, Madrid